CLINICAL TRIAL: NCT01957241
Title: Serum Biomarker Study for the Prognosis of Patients With Hepatocellular Carcinoma and Esophageal Cancer Undergoing Radiotherapy Using Multiplex Proximity Ligation Assay
Brief Title: PLA for HCC and Esophageal ca Serum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20110606IRC
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Hepatocellular Carcinoma; Esophageal Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We have collected the serum samples of patients before, during, and after RT with consent of two completed clinical trials and one active trial.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatocellular Carcinoma and Esophageal Cancer

SUMMARY:
The primary goal of this study is to quantify the biomarkers of pre-radiation therapy(RT), during-RT, and post-RT serum samples from hepatocellular carcinoma (HCC) and esophageal cancer patients undergoing definitive or neoadjuvant RT, and to correlate them with tumor response, patterns of failure, survival outcome, and RT-related lung or liver toxicity. The secondary goal of this study is to set up the PLA platform in our institute for future biomarker test.

DETAILED DESCRIPTION:
There have been many biomarkers, such as angiogenesis factors and cytokines, related to cancer progression or microenvironment interaction. However, the commonly used enzyme-linked immunosorbent assay (ELISA) requires the certain volume of each sample for specific antigen or antibody. It may not be practically efficient to test a broad spectrum of biomarkers with limited volumes of serum from cancer patients. Proximity ligation assay (PLA), an established concept and platform requiring very little sample volume to quantitatively detect a variety of biomarkers, is being developed with multiplex versions of improved sensitivity and dynamic range by the Stanford group. From the three completed trials ("In vivo/vitro radiation-induced liver disease in HBV carrier（9261700196）", "Bystander effect study of radiation-induced viral hepatitis B reactivation（9261700196）", and "Pre- and post-chemoradiation blood RNA-microarray analysis to predict response and outcome of locally advanced esophageal squamous cell carcinoma（200805061R）") and one ongoing trial ("A phase I dose escalation trial of conformal hypofractionated radiation therapy for patients with hepatitis B virus-related Child A cirrhosis and hepatocellular carcinoma（200906051R）"), we have collected the pre-treatment and post-treatment serum samples of patients with hepatocellular carcinoma undergoing definitive radiotherapy and patients with esophageal cancer undergoing neoadjuvant chemoradiotherapy. Altered patterns of failure for post-radiotherapy hepatocellular carcinoma, especially intrahepatic and extrahepatic metastasis, and treatment response for post-chemoradiotherapy esophageal cancer upon esophagectomy, demands the effective biomarkers for the early prediction and appropriate management. The limited sample volumes form the obstacle of testing adequate number of biomarkers by ELISA. In this study we plan to collaborate with the Stanford group, to send and process these samples (100 μL each) to measure the dynamic changes of up to 56 or more biomarkers. We try to find the potential biomarkers correlating with treatment responses and patterns of failure for the future clinical practice, and wish to set up this viable PLA platform in our institute through this collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of locally advanced esophageal cancer or Hepatocellular Carcinoma, RT is indicated
* Informed consent signed

Exclusion Criteria:

* not completed RT

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We collected the pre-treatment and post-treatment serum samples of patients with hepatocellular carcinoma undergoing definitive radiotherapy and patients with esophageal cancer undergoing neoadjuvant chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
BIOMARKER PANEL SELECTION AND MODELING | 3 years
  All statistical analyses completed in this study are executed using the R statistical computing environment. To select the discrete set of biomarkers used to fit models of HCC or esophageal cancer diagnosis, we use the R distribution of the Prediction Analysis of Microarrays statistical technique, PAMR. Logistic regression models are fit using the generalized linear model function in R.

SECONDARY OUTCOMES:
SURVIVAL AND RT-RELATED TOXICITY ANALYSIS AND MODELING | 3 years
  Survival data are fit to a right-censored model using the Survival function in the R statistical computing environment. Univariate and multivariate Cox proportional hazards models are fit onto survival data using the coxph function. Hazard ratios are calculated as the ratios of risk by the increase or decrease of 1 log2 PLA unit (2-fold increase or decrease in serum concentration of a biomarker). Lung or liver toxicity is graded by Common Toxicity Criteria version 3.0. Grade of toxicity is defined as the categorical variable and is correlated with the ratios of risk by the increase or decrease of 1 log2 PLA unit.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chia-Hsien Cheng, MD, PhD, Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan